CLINICAL TRIAL: NCT05913453
Title: Technical Failure During Colorectal Endoscopic Full Thickness Resection (EFTR): The "Through Thick and Thin" Study
Status: Completed | Type: Observational
Sponsor: Azienda Unità Sanitaria Locale della Romagna (Other)
Responsible Party: Principal Investigator, Carlo Fabbri, Dr., Azienda Unità Sanitaria Locale della Romagna
Other Study IDs: 2993
Record Dates: First submitted 2023-03-24; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Endoscopic Full Thickness Resection (EFTR); Residual /Recurrent Colorectal Lesion; Full-thickness Resection Device (FTRD); Colorectal Adenoma; Non-lifting Colorectal Lesions; Intraprocedural Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Procedures corresponding to technical failure

SUMMARY:
Among advanced resection techniques, endoscopic full thickness resection (EFTR) allows closure and full-thickness resection by the use of the non-exposed full thickness resection device (FTRD). The study is a retrospective analysis of technical failure occurring during colorectal full-thickness resection. Full thickness resection is a safe and effective procedure for "difficult" colorectal lesions. However, technical failure can occur and to date there is no evidence about type and clinical consequences in this setting.

DETAILED DESCRIPTION:
The study is a multicentre retrospective study involving centres with experience in advanced colorectal resections.

Each centre is invited to submit information about the Centre and to report alle the consecutive cases corresponding to technical failure.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive colorectal EFTR procedures with technical failure by using OVESCO Full Thickness Resection Device

Exclusion Criteria:

* EFTR performed by exposed techniques and/or devices different from FTRD
* Patients not able to give informed consent for data collection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colorectal EFTR with occurrence of technical failure.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Technical failure rate and classification | 2014 - 2022

SECONDARY OUTCOMES:
Conservative Management of technical failure | 2014-2022
  Performance of rescue endoscopic resection
Clinical success (R0 resection) | 2014-2022
Complication rate | 2014-2022

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Morgagni-Pierantoni, Forlì, Forlì-Cesena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data require data about experience in colorectal resections and EFTR; each centre will provide details for each technical failure including demographics, lesions characteristics, intraprocedural details and post-procedure outcomes.

REFERENCES:
- [Derived] Gibiino G, Binda C, Papparella LG, Spada C, Andrisani G, Di Matteo FM, Gagliardi M, Maurano A, Sferrazza S, Azzolini F, Grande G, de Nucci G, Cesaro P, Aragona G, Cennamo V, Fusaroli P, Staiano T, Soriani P, Campanale M, Di Mitri R, Pugliese F, Anderloni A, Cucchetti A, Repici A, Fabbri C; "through thick and thin" study group. Technical failure during colorectal endoscopic full-thickness resection: the "through thick and thin" study. Endoscopy. 2024 Nov;56(11):831-839. doi: 10.1055/a-2328-4753. Epub 2024 May 16. PMID 38754466